CLINICAL TRIAL: NCT05078840
Title: Treatment of Patients With Diffuse Large B-cell Non-Hodgkins Lymphoma in Stages I and II Without Risk Factors, Adapted to the Response Evaluated With PET CT (Positron Emission Computed Tomography)
Brief Title: PET Adapted Treatment of Patients With Limited Stage DLBCL and no Risk Factors
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Grupo Argentino de Tratamiento de la Leucemia Aguda (Other)
Responsible Party: Sponsor
Other Study IDs: GATLA 10-LNHDCG-20
Record Dates: First submitted 2021-09-21; First posted 2021-10-15 (Actual); Last update posted 2024-01-09 (Actual); Status verified 2024-01

CONDITIONS: Lymphoma, Non-Hodgkin's, Adult
Keywords: PET; DLBCL
MeSH Terms: conditions — Lymphoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 36 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with DLBCL limited stages and without risk factors: Patients with DLBCL in limited stages and without risk factors that will receive standard chemoimmunotherapy and their treatment will be adapted according to PET response after 3 cycles.
  Interventions: Other: Evaluation of first line treatment in patients with stage I and II LBCL

INTERVENTIONS:
Other: Evaluation of first line treatment in patients with stage I and II LBCL — Evaluation of first line treatment in patients with stage I and II LBCL, without poor prognostic factors with treatment adapted to PET-CT after 3 R-CHOP

SUMMARY:
Prospective, multicenter, phase IV study, of real-life evidence destined to evaluate the feasibility and efficacy of performing a treatment adapted to PET-CT in patients with stage I and II DLBCL, without poor prognostic factors.

DETAILED DESCRIPTION:
Patients older than 17 years of age, with no upper age limit with a de novo histological diagnosis of DLBCL, in stages I and II and without risk factors, will be included. All patients will have a baseline PET-CT and will undergo 3 cycles of R-CHOP (cyclophosphamide, doxorubicin, vincristine, prednisone). A PET-CT will be performed on day 15-18 of the third cycle that will be centrally reviewed. Those patients with negative PET-CT (Deauville 1, 2 and 3) will receive an additional cycle of R-CHOP and will finish treatment. Patients who have PET-CT with a Deauville 4 score will complete a fourth cycle and then receive radiation therapy to the compromised site. Those patients with a Deauville score of 5 should receive rescue therapy, so they will be outside the protocol.

A standardized follow-up of the patients included with tomographic controls will be carried out, evaluating OS (overall survival) and PFS (progression-free survival) at 3 years as the main objectives.

ELIGIBILITY:
Inclusion Criteria:

* Patients > 17 years old with no upper age limit.
* Histological diagnosis of DLBCL Stages I or II
* Patients who have signed informed consent.

Exclusion Criteria:

* Patients with elevated LDH (lactate dehydrogenase)
* ECOG (Eastern Cooperative Oncology Group) > 2
* Stage III or IV
* Bulky mass (> 7.5 cm)
* Central nervous system involvement
* Testicular lymphoma
* Breast involvement
* Eyeball involvement
* Primary mediastinal lymphoma
* Cutaneous primary lymphoma
* Diffuse large B-cell lymphoma of the leg
* HIV positive patients
* Platelet count <100,000 / mcl and total leukocyte count <3,000 / mcl
* Marked impairment of ventricular function (FEy <50%)
* Moderate / severe renal impairment defined by Cl. Cr. <50 ml / min
* Severe liver disease: prothrombin rate <50% and / or bile level. total> 2.5 times normal value
* Pregnant and breastfeeding
* Previous or concomitant diagnosis of indolent lymphoma
* Patients who have previously received chemotherapy and / or radiotherapy

Min Age: 17 Years | Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: Adult patients with recent diagnosis of DLBCL in limited stages without risk factors and no previous history of mliagnant disease.
Sampling Method: Non-Probability Sample
Enrollment: 75 (Estimated)
Dates: Start 2021-06-01 (Actual); Primary Completion 2024-06-01 (Estimated); Study Completion 2025-06-01 (Estimated)

PRIMARY OUTCOMES:
Evaluate PFS in patients with stage I and II LBCL (large B cell lymphoma), without poor prognostic factors with treatment adapted to PET-CT after 3 R-CHOP. | 36 months
Evaluate OS in patients with stage I and II LBCL, without poor prognostic factors with treatment adapted to PET-CT after 3 R-CHOP | 36 months

SECONDARY OUTCOMES:
Evaluate PFS in patients with negative PET after 3rd cycle who shortened treatment to only 4 cycles of R-CHOP. | 36 months
Evaluate PFS in patients with positive PET after 3rd cycle who continue treatment with R-CHOP x 1 and Radiotherapy. | 36 months
Evaluate the prognostic value of baseline MTV (metabolic tumor volume) in patients with DLBCL under treatment adapted to response after 3 cycles of R-CHOP | 36 months
Evaluate the prognostic value of baseline TLG (total lesion glycolysis) in patients with DLBCL under treatment adapted to response after 3 cycles of R-CHOP | 36 months
Evaluate the prognostic value of Δ SUV (standardized uptake value) max in interim PET in patients with DLBCL under treatment adapted to response after 3 cycles of R-CHOP | 36 months
Compare our results in terms of OS and PFS with those described in patients treated with R-CHOP x6 | 36 months
Compare our results in terms of OS and PFS with those described in patients with treatments adapted to the result of PETi (interim PET) with R-CHOP x 4 (4 cycles of CHOP) | 36 months
Compare our results in terms of OS and PFS with those described in patients with treatments adapted to the result of PETi with R-CHOPx4+ 2 Rituximab or R-CHOPx 4 + ISRT (involved site radiation therapy) + Zevalin | 36 months
Compare our results in terms of OS and PFS with those described in patients with treatments adapted to the result of PETi with R-CHOPx 4 + RTCC + Zevalin | 36 months

CONTACTS AND LOCATIONS:
Overall Officials: Amalia Cerutti, Dr., Principal Investigator — Grupo Argentino de Tratamiento de la Leucemia Aguda; Astrid Pavlovsky, Dr., Study Chair — Grupo Argentino de Tratamiento de la Leucemia Aguda
Locations (7):
- Argentina (7):
  - Hospital Italiano de La Plata, La Plata, Buenos Aires
  - Instituto Privado de Hematologia y Hemoterapia, Paraná, Entre Ríos Province
  - IDHEA Clínica Hematológica, Rosario, Santa Fe Province
  - FUNDALEU, CABA
  - Hospital Italiano de Buenos Aires, CABA
  - Clínica Universitaria Reina Fabiola, Córdoba
  - Hospital Privado de Córdoba, Córdoba

IPD SHARING:
Plan to Share IPD: Yes
Share study protocol
Supporting Information: Study Protocol
Time Frame: The data will become available on June 2021, and will remain available until the end of the clinical trial.